CLINICAL TRIAL: NCT02219295
Title: Sensory and Gastrointestinal Impact of Taste Receptor Variants on Human Metabolism and Nutrition
Brief Title: SEGATROM: Sensory and Gastrointestinal Impact of Taste Receptor Variants on Human Metabolism and Nutrition
Acronym: SEGATROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Prof. Dr. med., German Institute of Human Nutrition
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: BMBF 11005D
Record Dates: First submitted 2014-08-01; First posted 2014-08-18 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Disorder of Glucose Regulation
Keywords: SGLT1 (sodium dependent glucose transporter); Glut-transporters; taste receptors genes; sweet taste receptor T1R2T1R3; bitter taste receptors of the hTAS2gene family
MeSH Terms: interventions — Sugars; Sucrose; Glucose; isomaltulose; Galactose; Sweetening Agents; Saccharin; sinigrin; intybin; oxytocin, 1-alpha-mercaptoacetic acid-iso-Asn(5)-; Gastroscopy; Sodium-Glucose Transporter 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- sweet -block (Experimental): application of different sugars, artificial sweeteners and sweet-taste antagonists in a single dose in 300 ml tap water every week up to 7 times and collection of blood samples over 3 hours
  Interventions: Dietary Supplement: sweet block; Dietary Supplement: bitter block; Dietary Supplement: umami-block
- bitter block (Experimental): application of purified bitter tasting ingredients of vegetables and hop in 300 ml tap water , collection of blood samples for 3h (-15,0,15,30,60,120,180 min)
  Interventions: Dietary Supplement: sweet block; Dietary Supplement: bitter block; Dietary Supplement: umami-block
- umami-block (Experimental): application of glutamate and glutamate +IMP
  same procedure as above
  Interventions: Dietary Supplement: sweet block; Dietary Supplement: bitter block; Dietary Supplement: umami-block
- gastroscopy (Other): gastroscopy with and without oral intervention with artificial sweetener saccharin to take tissue samples from the upper bowel for the investigation of taste receptor cells in the upper bowel in human beings
  Interventions: Other: gastroscopy

INTERVENTIONS:
Dietary Supplement: sweet block — oral application of the above mentioned substances in 300 ml tap water in 5 min. , collection of blood at 0,15,30, 60 ,120,180 minutes for measurement of incretins GIP(gastrointestinal polypeptide) and GLP-1 (glucagon like peptide 1), Protein hormones PYY(Peptide YY),CCK (cholecystokinin), Leptin and Insulin
  Other Names: Sugars as sucrose, glucose, palatinose, galactose; artificial sweeteners as saccharin; sweet taste antagonist as lactisol
  Arms: bitter block; sweet -block; umami-block
Dietary Supplement: bitter block — oral application of the above mentioned substances in 300 ml tap water, collection of blood samples at -15,0,15,30,60,120,180 min for Insulin, GIP,GLP-1, PYY and glucose
  Other Names: application of; sinigrin; lactucopicrin; iso-alpha-acid
  Arms: bitter block; sweet -block; umami-block
Dietary Supplement: umami-block — oral application of umami substances as glutamate with and without IMP, collection of blood samples as above
  Other Names: application of glutamate and glutamate+IMP,
  Arms: bitter block; sweet -block; umami-block
Other: gastroscopy — gastroscopy with and without oral application of saccharin, tissue samples from th upper duodenum by endoscopy for the detection of taste receptor cells in the upper bowel
  Other Names: tissue samples; sweet taste receptor stimualtion; artificial sweetener saccharin; SGLT-1
  Arms: gastroscopy

SUMMARY:
We investigate the impact of taste receptors (sweet, bitter and umami) on human metabolism. There ist growing evidence, that components of the taste signalling system, including the taste receptor proteins , have important functions in the regulation of metabolic parameters in non-gustatory tissues.

DETAILED DESCRIPTION:
We apply different sweet, bitter and umami taste compounds in a single dose in the human intervention. We use substances as for instance glucose, sucrose,saccharin and lactisol in the sweet part, and substances from cabbage, beer or red endive in the bitter part. For umami we take glutamate.

Blood samples are collected at baseline and 6 times thereafter up to 3hours, to analyse the incretins GLP-1(glucagon-like peptide 1) and GIP(gastrointestinal polypeptide) and other peptide hormones as insulin and PYY(peptide tyrosin trosin) in human beings.

Gastrointestinal mucosa is taken by gastroscopy from the lower duodenum from study subjects for analysis for the presence or absence of functional taste receptors in gastrointestinal tissues.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons

Exclusion Criteria:

* Tumor in history
* Pregnancy
* Severe illness in history
* Bodymass index below 18

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC): changes of expression levels of the sweet , bitter und umami taste receptors in humans in the upper bowel and responses of incretins to receptor agonists and antagonists | three years
  measurement of incretins (GIP, GLP-1) and peptide hormones in human plasma after consumption of different sugars , sweeteners , bitter tasting ingredients of vegetables und umami. Measurement of expression levels in human intestinal mucosa before and after receptor stimulation

SECONDARY OUTCOMES:
changes in the signalling cascade of the sweet receptor SGLT1 (sodium tranporter 1), changes of receptor expression | 3 years
  oral application of sweet tasting substances and antagonists, endoscopic collection of tissue samples, determination of molecular resonses by qRT-PCR and immunohistochemistry

OTHER OUTCOMES:
Changes in the Area under the Curve (AUC) for PYY in different bitter tasting substances | 3 years
  oral application of sinigrin, lactucopicrin and other extracts of vegetables and umami, getting insight into the different bitter receptors

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Peiffer, Prof, Principal Investigator — German Institute of Human Nutrition
Locations (1):
- Department of Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg, Germany

REFERENCES:
- [Derived] Zhang J, Schafer SM, Kabisch S, Csanalosi M, Schuppelius B, Kemper M, Markova M, Meyer NMT, Pivovarova-Ramich O, Keyhani-Nejad F, Rohn S, Pfeiffer AFH. Implication of sugar, protein and incretins in excessive glucagon secretion in type 2 diabetes after mixed meals. Clin Nutr. 2023 Apr;42(4):467-476. doi: 10.1016/j.clnu.2023.02.011. Epub 2023 Feb 21. PMID 36857956
- [Derived] Keyhani-Nejad F, Kemper M, Schueler R, Pivovarova O, Rudovich N, Pfeiffer AF. Effects of Palatinose and Sucrose Intake on Glucose Metabolism and Incretin Secretion in Subjects With Type 2 Diabetes. Diabetes Care. 2016 Mar;39(3):e38-9. doi: 10.2337/dc15-1891. Epub 2015 Dec 30. No abstract available. PMID 26721819